CLINICAL TRIAL: NCT01381380
Title: Effect of Manual Therapy After Trigger Point Injection for Myofascial Pain Syndrome
Brief Title: Manual Therapy Treatment for Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Rioko Kimiko Sakata, Universidade Federal de São Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1276
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-11

CONDITIONS: Myofascial Pain Syndromes
Keywords: myofascial pain; trigger point injection; manual therapy
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Musculoskeletal Manipulations; Massage; Myofascial Release Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm studies (Other): Manual therapy for one group
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Procedure: Manual therapy — Manual therapy, once a week for 8 weeks
  Other Names: massage; finger pressure; myofascial release; mobilization

SUMMARY:
This study is a pain intensity evaluation in patients with myofascial pain submitted kinesitherapy after trigger point injection.

DETAILED DESCRIPTION:
Randomized prospective study conducted on 30 patients of both genders ranging in age from 18 to 60 years, with neck and shoulder girdle Myofascial Pain Syndrome (MFS), with a duration of ≥ 4 months and pain intensity ≥ 4.

Trigger point injection of 1 mL 0.25% bupivacaine at each point, once a week for 8 weeks (T1 to T8).

Group 1: kinesiotherapy once a week for 8 weeks Group 2: not submitted to kinesiotherapy Evaluation of pain intensity on the first assessment (T0) and after 1, 2, 3, 4, 5, 6, 7, 8, and 9 weeks

ELIGIBILITY:
Inclusion Criteria:

* myofascial pain of neck and shoulder girdle, lasting ≥ 4 months, pain intensity ≥ 4.

Exclusion Criteria:

* arrhythmia
* heart block
* coagulopathy
* cognitive alterations and infection at the site
* patients using anticoagulants, and pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks
  once a week for 8 weeks (T1 to T8)

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, PhD, Study Director — Universidade Federal de São Paulo
Locations (1):
- Setor de Dor, São Paulo, São Paulo, Brazil